CLINICAL TRIAL: NCT01168531
Title: The Effect of Pregabalin and Dexamethasone on Acute and Chronic Pain After Lumbar Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Jae Kwang Shim / Assistant Professor, Department of Anesthesiology & Pain Medicine, Severance Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2009-0506
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-01

CONDITIONS: Pain
Keywords: patients undergoing lumbar spinal surgery
MeSH Terms: conditions — Pain | interventions — Pregabalin; Dexamethasone

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo arm (Placebo Comparator)
  Interventions: Drug: placebo
- pregabalin arm (Active Comparator)
  Interventions: Drug: Pregabalin
- dexamethasone with pregabalin arm (Experimental)
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: Pregabalin — pregabalin: 300 mg/day, po, from operative day until third postoperative day.
  Arms: pregabalin arm
Drug: dexamethasone — Dexamethasone 16 mg, intravenous, before induction of anesthesia
  Arms: dexamethasone with pregabalin arm
Drug: placebo — vitamin B complex formula
  Arms: placebo arm

SUMMARY:
Multimodal analgesia may be important for optimal postoperative pain treatment and facilitation of early mobilization and recovery. This study investigated the analgesic effect of pregabalin and dexamethasone in patients undergoing lumbar spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for lumbar spinal surgery, aged 20 to 70 years, with a body mass index (BMI) from 18 to 32 and an American Society of Anesthesiologists (ASA)physical status classification of I-II were eligible for the study.

Exclusion Criteria:

* allergy to any drugs in the study
* alcohol and/or drug abuse
* treatment with antacids or antidepressants
* a history of diabetes or epilepsy
* a daily intake of analgesics or an intake of any analgesic within 24 h before surgery
* treatment with systemic glucocorticoids within 4 weeks before surgery
* known impaired hepatic and renal function.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
the multimodal analgesic effect of pregabalin, and of pregabalin with dexamethasone | Assessment was performed during the first 72 hour following emergence from general anesthesia, subdivided into 5 time periods; on arrival of patient to the PACU, 1-6 hour, 6-24 hour, 24-48 hour and 48-72 hour
  Primary Outcome is to investigate the multimodal analgesic effect of pregabalin, and of pregabalin with dexamethasone, in patients receiving a patient-controlled analgeisa with fentanyl, on fentanyl consumption (primary end point), pain scores and side effects in patients scheduled for lumbar spinal surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea